CLINICAL TRIAL: NCT04096859
Title: Assessment of PremiCron Suture for Cardiac Valve Reconstruction and Replacement. A Multi-centric, Prospective, Single Arm Observational Study in Daily Practice.
Brief Title: PremiCron Suture for Cardiac Valve Repair
Acronym: PremiValve
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Collaborators: B.Braun Surgical SA (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1823
Record Dates: First submitted 2019-09-18; First posted 2019-09-20 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Aortic Valve Stenosis
Keywords: elective surgery; minimally invasive surgery; cardiac valve reconstruction; cardiac valve replacement
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PremiCron®: Assessment of PremiCron suture for cardiac valve reconstruction and replacement

SUMMARY:
The study is a voluntary study, initiated by B. Braun to collect clinical data for PremiCron® suture concerning its key indication.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing an elective primary open or minimal invasive surgery for a single or multiple cardiac valve reconstruction or / and replacement.
* Age ≥18 years
* Written informed consent

Exclusion Criteria:

* Patients undergoing an elective primary cardiac valve reconstruction or / and replacement in combination with a coronary arterial bypass graft surgery.
* Emergency surgery
* Pregnancy
* Infective endocarditis
* Previous cardiac surgical intervention
* Known immunodeficiency or immunosuppression
* Participation or planned participation in another cardiovascular study before study follow-up is completed.
* Inability to give informed consent due to mental condition, mental retardation, or language barrier.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients
Sampling Method: Non-Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2019-11-22 (Actual); Primary Completion 2021-09-02 (Actual); Study Completion 2022-01-13 (Actual)

PRIMARY OUTCOMES:
a composite endpoint of Myocardial infarction, Stroke, Mortality until discharge and rate of Endocarditis of the replaced / reconstructed valve until 6 months | from intervention up to 6 months postoperative
  a composite endpoint of
  * Myocardial infarction until discharge
  * Stroke until discharge
  * Mortality until discharge
  * Endocarditis of the replaced / reconstructed valve until 6 months

SECONDARY OUTCOMES:
Comparison of mortality at different timepoints in postoperative course | until discharge (approximately 10 days postoperative), 30 days and 6 months postop
  Incidence of mortality until discharge, 30 days and 6 months postop
Comparison of myocardial infarction (MI) at different timepoints in postoperative course | until discharge (approximately 10 days postoperative), 30 days and 6 months postop
  Incidence of myocardial infarction (MI) until discharge, 30 days and 6 months postop
Comparison of stroke at different timepoints in postoperative course | until discharge (approximately 10 days postoperative), 30 days and 6 months postop
  Incidence of stroke until discharge, 30 days and 6 months postop
Comparison of endocarditis of the replaced / reconstructed valve at different timepoints in postoperative course | until discharge (approximately 10 days postoperative), 30 days and 6 months postop
  Incidence of endocarditis of the replaced / reconstructed valve until discharge, 30 days and 6 months postop
Comparison of superficial and deep chest wound infections valve at different timepoints in postoperative course | until discharge (approximately 10 days postoperative), 30 days and 6 months postop
  Incidence of superficial and deep chest wound infections until discharge, 30 days and 6 months postop
Comparison of atrial fibrillation valve at different timepoints in postoperative course | until discharge (approximately 10 days postoperative), 30 days and 6 months postop
  Incidence of atrial fibrillation until discharge, 30 days and 6 months postop
Comparison of renal failure at different timepoints in postoperative course | until discharge (approximately 10 days postoperative), 30 days and 6 months postop
  Incidence of renal failure until discharge, 30 days and 6 months postop
Comparison of pneumonia at different timepoints in postoperative course | until discharge (approximately 10 days postoperative), 30 days and 6 months postop
  Incidence of pneumonia until discharge, 30 days and 6 months postop
Comparison of mediastinitis at different timepoints in postoperative course | until discharge (approximately 10 days postoperative), 30 days and 6 months postop
  Incidence of mediastinitis until discharge, 30 days and 6 months postop
Comparison of bleeding at different timepoints in postoperative course | until discharge (approximately 10 days postoperative), 30 days and 6 months postop
  Incidence of bleeding until discharge, 30 days and 6 months postop
Rate of adverse events | until 6 months postop
  valve related reoperation, haemothorax, paravalvular leak, pacemaker insertion, embolism, valve insufficiency, gastrointestinal bleeding, surgery not valve related
Length of intensive care unit stay | until discharge (approximately 10 days postoperative)
  Number of days the patient has to stay in intensive care unit after intervention
Length of hospital stay | until discharge (approximately 10 days postoperative)
  Number of days the patient has to stay in hospital
Intraoperative handling of the suture material | intraoperative
  Intraoperative handling of the suture material using a questionnaire containing different dimension and a 5 point assessment level (Likert Scale), including pledget assessment
Course of Health Status | until 6 months postoperative
  EQ-5D is a standardized measure of health status developed by EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal. EQ-5D is designed for self-completion by respondents and it takes only a few minutes to complete. Instructions to respondents are included in the questionnaire. EQ-5D-5L consists of 2 pages - descriptive system and the EQ visual Analogue scale (EQ-VAS). The descriptive system comprises 5 dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression). Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The EQ VAS records the respondents self rated health on a 20 cm vertical , visual analogue scale with endpoints labelled "the best health you can imagine" and " the worst health you can imagine"
Employment status | preoperative and 6 months postoperative
  The employment status of the patient before / after the intervention to evaluate the influence of cardiac valve reconstruction or / and replacement on employment

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich FW Franke, Prof. Dr. med., Principal Investigator — Robert Bosch KrankenhausDepartment for Thoracic and Vascular Surgery
Locations (2):
- Robert Bosch KH Stuttgart, Stuttgart, Germany
- Hospital de la Santa Creu I Sant Pau, Barcelona, Spain

REFERENCES:
- [Result] Rufa M, Ursulescu A, Baumann P, Ferrer MT. A prospective, international, bicentric study to evaluate PremiCron suture material for cardiac valve surgery - PREMIVALVE a cohort study. Ann Med Surg (Lond). 2023 Apr 4;85(4):835-841. doi: 10.1097/MS9.0000000000000442. eCollection 2023 Apr. PMID 37113912